CLINICAL TRIAL: NCT00692627
Title: Evaluation of Volume Status, Haemodynamics and Microcirculatory Flow in Adult Patients With Severe Falciparum Malaria
Acronym: PRiSM
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Josh Hanson, Mahidol Oxford Research Unit
Other Study IDs: BKMAL0804
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Severe Falciparum Malaria
Keywords: Falciparum; malaria; volume; haemodynamics
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
acidosis, acute renal failure and acute pulmonary oedema are common, and frequently fatal, manifestations of severe P. falciparum malaria. The course of all three might be ameliorated by optimising a patient's intravenous fluid therapy. The fluid treatment of severe malaria is presently empirical, by defining cardiovascular responses to volume replacement we would provide a physiological basis for resuscitation strategies.

We will use pulse contour cardiac output monitoring (PiCCOTM) to guide the fluid resuscitation of patients admitted to intensive care with severe malaria. With data collected during the patients' admission we hope to:

1. Assess the degree of hypovolaemia in adults with severe malaria and its contribution to microcirculatory dysfunction and acidosis.
2. To assess the relationships between volume status, haemodynamic parameters and the renal and pulmonary manifestations of severe malaria.
3. To assess the utility of central venous pressure measurement as a guide for fluid administration in patients with severe malaria
4. To investigate the prognostic and clinical utility of central venous oxygen saturation in severe malaria

In this way we hope to develop a greater understanding of the pathophysiology of haemodynamic derangement in severe malaria. By comparing the PiCCO derived data with simpler clinical parameters, we hope to determine potential fluid resuscitation strategies - relevant for a resource poor setting - whose efficacy could be confirmed in future trials.

ELIGIBILITY:
Inclusion Criteria

1. Severe malaria, defined by the modified criteria of Hien et al and the presence of asexual forms of P. falciparum in the peripheral blood smear.
2. The patients or their attending relative able and willing to give fully informed written consent.
3. Age ≥ 16 years

Exclusion Criteria

1. Patients or relatives unable or unwilling to give informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe Falciparum Malaria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Metabolic Acidosis | 48 hours

SECONDARY OUTCOMES:
Acute renal failure | By discharge
Acute pulmonary oedema | By discharge

CONTACTS AND LOCATIONS:
Overall Officials: Arjen Dondorp, MD, Study Director — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh

REFERENCES:
- [Derived] Hanson J, Lam SW, Alam S, Pattnaik R, Mahanta KC, Uddin Hasan M, Mohanty S, Mishra S, Cohen S, Day N, White N, Dondorp A. The reliability of the physical examination to guide fluid therapy in adults with severe falciparum malaria: an observational study. Malar J. 2013 Oct 1;12:348. doi: 10.1186/1475-2875-12-348. PMID 24079262